CLINICAL TRIAL: NCT03447106
Title: An Analysis of Costs and Outcomes Based on the Open, Laparoscopic, and Da Vinci Robotic Approach for Gastric Cancer Resection.
Brief Title: Comparison of Open Laparoscopic and Robotic Surgery in Gastric Cancer Resection.
Acronym: Cooladvrsigcr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2018-001
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Laparotomy; Laparoscopy; Robotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open (Experimental)
  Interventions: Procedure: laparotomy
- Laparoscopic (Experimental)
  Interventions: Procedure: Laparoscopic
- Robotic (Experimental)
  Interventions: Procedure: Robotic

INTERVENTIONS:
Procedure: laparotomy — This is a kind of traditional surgical method.
  Arms: Open
Procedure: Laparoscopic — laparoscopic surgery
  Arms: Laparoscopic
Procedure: Robotic — the Da Vinci robot assisted gastric resection
  Arms: Robotic

SUMMARY:
Gastric cancer is a common gastrointestinal tumor, and surgical operation is still the main method of gastric cancer treatment. Reported for the first time since 1994, the laparoscopic gastric cancer radical prostatectomy, laparoscopic technique is widely applied in the field of gastrointestinal surgery, has gradually replaced the traditional open operation as the main mode of surgical treatment for gastric cancer. Although laparoscopy has many advantages, there are still disadvantages, such as the discomfort of the physician, the reverse operation, and the ease of shaking, which hinder the application of laparoscopy. In recent years, the Da Vinci robot assisted gastric resection has become a new way to treat gastric cancer. Compared with the traditional laparoscopy and laparotomy, the operation of the robot is more precise and flexible, with obvious advantages of minimally invasive and good application value and prospect. The aim of the study is to compare value (outcomes/costs) of surgery in patients with Gastric Cancer by 3 approaches: open, laparoscopic, and robotic.First of all, the investigators will collect 500 cases of Gastric Cancer patients, randomly assigned for the open, laparoscopic, and robotic group. Secondly, to analyzing the demographic data,basic treatment and follow-up data, including the operation time, blood loss, the number of cut edge positive, the distances of cut edge away from the tumor edge, the cases of anastomotic fistula bleeding, stenosis, average such confinement, the meal time, cost of treatment, tumor recurrence rate, the presence of residual stomach, upset stomach and frequency, reflux esophagitis, bile reflux gastritis and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients without contraindications gastroscope，surgery and anesthesia;
* There is no history of abdominal surgery, no severe abdominal cavity adhesion
* Patients signed informed consent

Exclusion Criteria:

* Patients with preoperative assessment of distant metastasis;
* Patients with preoperative radiation and chemotherapy or hormone therapy;
* Patients with acute obstruction, bleeding or perforation of the emergency surgery
* Patients with a history of abdominal trauma or abdominal surgery.
* Patients with contraindications gastroscope，surgery and anesthesia;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence rate | 2 years
cost of treatment | 2 years

SECONDARY OUTCOMES:
the operation time | one hour-six hours

OTHER OUTCOMES:
the all number of postoperative complications（ frequency,reflux esophagitis and bile reflux gastritis） | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jun She, M.D; PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China